CLINICAL TRIAL: NCT05077462
Title: An Open Label, Randomized, Single Dose, 2-sequence, 2-period, Cross-over Phase 1 Study to Evaluate the Safety and Pharmacokinetics of AJU-C52H Compared to Coadministration of C52R1M With C52R2 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Evaluate the Safety and Pharmacokinetics of AJU-C52H in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21HT10602
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: C52R1M(Valsartan/Amlodipine) and C52R2(Chlorthalidone), single dose Period 2: AJU-C52H(FDC tablet, Valsartan/Amlodipine/Chlorthalidone), single dose
  Interventions: Drug: C52R1M Tab. and C52R2 Tab.; Drug: AJU-C52H
- Sequence B (Experimental): Period 1: AJU-C52H(FDC tablet, Valsartan/Amlodipine/Chlorthalidone), single dose Period 2: C52R1M(Valsartan/Amlodipine) and C52R2(Chlorthalidone), single dose
  Interventions: Drug: C52R1M Tab. and C52R2 Tab.; Drug: AJU-C52H

INTERVENTIONS:
Drug: C52R1M Tab. and C52R2 Tab. — Single oral dose C52R1M(FDC, Valsartan/Amlodipine) 160/5 mg tablet and C52R2(Chlorthalidone) 25 mg tablet taken together
  Other Names: Reference Drug
Drug: AJU-C52H — Single oral dose AJU-C52(Valsartan/Amlodipine/Chlorthalidone) 160/5/25 mg FDC tablet
  Other Names: Test Drug

SUMMARY:
To evaluate the safety and pharmacokinetic characteristics of AJU-C52H in healthy adults

DETAILED DESCRIPTION:
This study is to assess the safety and pharmacokinetic characteristics between co-administration of C52R1M with C52R2 and administration of AJU-C52H.

This is an open-label, randomized, single-dose, 2x2 crossover study in healthy subjects to assess the bioequivalence after taking the study drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19-year-old
2. Weight ≥ 50kg (man) or 45kg (woman), with calculated body mass index(BMI) of 18 to 30 kg/m2
3. Those who are eligible for adequate blood pressure criteria during screening tests Systolic blood pressure: 90 to 139 mmHg Diastolic blood pressure: 60 to 89 mmHg
4. Those who have no congenital chronic disease or chronic disease requiring treatment and who have no pathological symptoms or findings
5. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serum, urine test) and 12-lead ECG results during screening tests
6. Those who agree to contraception during the participation of clinical trial
7. Those who voluntarily decide to participate and agree to comply with the cautions after hearing and fully understanding the detailed description of this clinical trial

Exclusion Criteria:

1. Those who received investigational product or bioequivalence test drug within 6 months before the first administration of clinical trial drug
2. Those who take barbiturate and related (causing induction or inhibition of metabolism) drug within 1 month before the first administration of clinical trial drug
3. Those who donated whole blood and apheresis within 8 weeks or received transfusion within 4 weeks
4. Those who has a history of gastrointestinal surgery
5. Those who exceeding an alcohol and smoke consumption criteria Alcohol: Men - 21 glass/week, Women - 14 glass/week (1 glass: Soju 50 mL, Beer 250mL, Wine 30 mL) Smoke: 20 cigarettes/day
6. Those who has a disease history of diabetic mellitus, nephropathy, biliary obstruction, dihydropyridine sensitivity, angioedema
7. Genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
8. Those who are deemed unfit by the investigators to participate in the clinical trial for other reasons including the results of laboratory tests
9. Women who are pregnant or who may be pregnant and breastfeed

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
AUCt of AJU-C52 | Pre-dose (0 hour), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  AUCt: Area under the concentration-time curve from time zero to time
Cmax of AJU-C52 | Pre-dose (0 hour), 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Cmax: Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, Republic of South Korea, South Korea